CLINICAL TRIAL: NCT05132335
Title: Assessment of Fatty Acid Uptake and Blood Flow in Tissues Under Fasting and Postprandial Conditions; a Repeatability Study Using Dynamic PET/MR Imaging in Patients With Type 2 Diabetes and Non-diabetic Control Subjects
Brief Title: A Repeatability Study of Fatty Acid Uptake Using PET/MR Imaging in Patients With T2DM and Non-diabetic Control Subjects
Acronym: AM05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Antaros Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AM05
Record Dates: First submitted 2021-10-29; First posted 2021-11-24 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: One arm: Subjects are studied under two consecutive conditions, after overnight fasting and after a liquid meal ingestion. During each condition they are examined for fatty acid uptake in subcutaneous fat and skeletal muscle by FTHA([18F]-FTHA) PET/MRI as well as adipose and skeletal muscle blood perfusion by radioactive water([15O]-H2O ) PET/MRI. This was done at two occasions, 2-14 days apart, to assess repeatability of the measurements.
  Assigned interventions:
  [18F]-FTHA tracer injections
  [15O]-H2O tracer injections
  PET/MRI imaging
  Overnight fasting Liquid meal ingestion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Imaging Biomarkers (Experimental): Each study subject is is studied in four session: twice after overnight fast and twice after liquid meal injestion using PETMRI imaging. Adipose and skeletal muscle pefusion and fatty adic uptake are measured and and the repeability of results tested for these two situations. In PEt studies PET/MRI Scan with radioactive water ([15O]-H2O) and [18F]-FTHA are used as tracers. In this experimental study number of subjects studied is rather small. Therefore volunteers with and without T2 diabetes are analysed together and not on different arms.
  Interventions: Other: Imaging Biomarkers

INTERVENTIONS:
Other: Imaging Biomarkers — One arm: Subjects are studied under two consecutive conditions, after overnight fasting and after a liquid meal ingestion. During each condition they are examined for fatty acid uptake in subcutaneous fat and skeletal muscle by FTHA([18F]-FTHA) PET/MRI as well as adipose and skeletal muscle blood perfusion by radioactive water([15O]-H2O ) PET/MRI. This was done at two occasions, 2-14 days apart, to assess repeatability of the measurements.
  Assigned interventions:
  [18F]-FTHA tracer injections [15O]-H2O tracer injections
  PET/MRI imaging
  Overnight fasting Liquid meal ingestion
  Other Names: Assessment of repeatability of fatty acid uptake in adipose using PETMRI

SUMMARY:
The main purpose of this study is to evaluate the overall variation in the assessment of fatty acid uptake and blood flow in adipose tissue and skeletal muscle in the fasted and postprandial states by evaluating the repeatability of whole-body three-dimensional kinetic (4D) combined positron emission tomography and magnetic resonance imaging (PET/MRI) readouts in participants with type 2 diabetes mellitus (T2DM), and non-diabetic control participants. Each volunteer participates 4 scanning sessions.

DETAILED DESCRIPTION:
A total of approximately 13 T2DM and 6 control subjects (a total of 19 subjects) are planned to be enrolled to achieve 11 T2DM and 5 control subjects to complete the study, assuming a 15% drop-out rate. The test-retest repeatability of the ratio of FTHA uptake rates in subcutaneous adipose tissue (SAT) to skeletal muscle is measured using the intra-class correlation coefficient (ICC). Assuming an ICC of 0.85, with a 5% two-sided type I error rate, a sample size of 16 completers will yield approximately 90% power to detect an ICC statistically significantly greater than 0.4 (usually considered as a criterion for moderate agreement).

The total radiaooin burden for tshi sitdu yis 27.4 mSv. The study is approved by the local Ethical committtee and Fimea.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 25 to 40 kilograms per meter squared (kg/m²),
* For participants with a confirmed type 2 diabetes diagnosis: The condition must be managed either by diet and exercise alone or on a stable dose of metformin
* For nondiabetic subjects: participants must agree to keep their diet and physical activity habits stable throughout the study
* Female participants must be post-menopausal and male participants

Exclusion Criteria:

* Poorly controlled diabetes
* Unstable body weight within 30 days prior to screening.
* For non-diabetic control subjects: evidence of diabetes or prediabetes at screening.
* Having worked as a metal worker or welder
* History of alcohol or drug abuse within 5 years of the screening
* Currently participating, or previous participation in another clinical trial within 30 days prior to the screening visit, or previous participation in another PET imaging study within 12 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the repeatability of the ratio of subcutaneous adipose tissue (SAT) to skeletal muscle fatty acid uptake rates | Baseline through Day 14
  The ratio of SAT to skeletal muscle fatty acid uptake rates

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo R Nuutila, MD, PhD, Principal Investigator — Turku PET Centre
Locations (2):
- Finland (2):
  - Turku PET Centre, Turku
  - Turku PET Centre (Turku University Hospital), Turku

IPD SHARING:
Plan to Share IPD: No
test-retest study, intermediate results not meaningful but the whole data set is reported.

REFERENCES:
- [Derived] Aarnio R, Kirjavainen A, Rajander J, Forsback S, Kalliokoski K, Nuutila P, Milicevic Z, Coskun T, Haupt A, Laitinen I, Haaparanta-Solin M. New improved radiometabolite analysis method for [18F]FTHA from human plasma: a test-retest study with postprandial and fasting state. EJNMMI Res. 2024 Jun 13;14(1):53. doi: 10.1186/s13550-024-01114-5. PMID 38869780